CLINICAL TRIAL: NCT06576128
Title: Analgesic Effect of Ultrasound-Guided Transversus Abdominis Plan (TAP) Block in Femoral Endovascular Cardiac Interventions: A Prospective-randomized Study
Brief Title: Ultrasound-Guided Transversus Abdominis Plan (TAP) Block in Endovascular Cardiac Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kerem Erkalp, MD, Prof, proffessor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-05

CONDITIONS: Anesthesiology; Percutaneous Coronary Intervention; Cardiac Catheterization; Analgesia; Satisfaction, Patient
Keywords: ultrasonography; anesthesiology; transversus abdominis plane block; Percutaneous Coronary Intervention; Cardiac Catheterization; analgesia
MeSH Terms: conditions — Agnosia; Patient Satisfaction | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Sham Comparator): only local anesthesia will be applied to surgical field as a part of the routine procedure.
  Interventions: Procedure: parenteral local anesthesia
- block group (Active Comparator): local anesthesia will be applied to surgical field as a part of the routine procedure and additionally transversus abdominisl plane block will be applied.
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — In additional to local anesthesia, 10 ml lidocaine (2%) (Lidon, Onfarma, Turkey ), TAPB will be performed under ultrasound imaging..
  Arms: block group
Procedure: parenteral local anesthesia — As routine procedure; the cardiologist will palpate the right or left femoral artery under sterile conditions and apply approximately 10 ml lidocaine (2%) to this area as local anesthesia (Lidon, Onfarma, Turkey ). Then, a puncture will be made on the anterior wall of the femoral artery with an 18 G needle . Approximately 3-4 mm skin incision will be made with the number 11 scalpel tip and the Seldinger technique will be continued. 6F femoral sheath to be placed, cardiac The catheterization process will begin.
  Arms: control group

SUMMARY:
Sensory innervation of the femoral region which is the entry point for endovascular cardiac interventions such as coronary angiography,cardiac catheterization and percutaneous coronary intervention is complex.It is thought that the ilioinguinal and iliohypogastric nerves contribute mostly.With transversus abdominis plane block(TAPB),it is planned to provide analgesia by creating a block in these nerve branches that contribute to the sensory innervation of the intervention area.In addition;it was aimed to investigate patient's and physician's satisfaction during the procedure.

DETAILED DESCRIPTION:
Cardiac catheterization was first performed by Werner Frossman in the late 1920s, when the ureteral catheter was advanced in the antecubital vein and demonstrated by fluoroscopy in the right atrium. Over the years, this method was developed; It has been used for more specific and complicated clinical situations.

Coronary angiography was first used for diagnostic purposes in the 1950s. It has continued to exist as a gold standard method in the diagnosis and treatment of coronary artery diseases and some other cardiac pathologies until today.

For endovascular cardiac interventions; femoral, brachial and radial arteries are used. Blood loss and difficulty in achieving hemostasis are harder in femoral artery interventions than other arteries. However, it has been observed that the femoral artery is more frequently preferred in endovascular cardiac interventions. The reason is that the artery has a large lumen (approximately 8-9 mm) and continues after the abdominal aorta and iliac artery. One of the most important reasons for this is that there is very little anatomical variation. The femoral artery can be felt approximately 1/3 medial to the inguinal ligament.After the inguinal ligament, the iliac artery, commonly it is called the femoral artery. Femoral artery is mostly preferred in cardiac interventions. Because this region has common iliac artery it is thought to be safer because it comes before the bifurcation of the femoral artery and after the inferior epigastric artery.

Transversus abdominis plane block (TAPB) aims to block the ilioinguinal and iliohypogastric nerves. In gynecological, urological surgeries, colorectal surgeries, cholecystectomies and inguinal surgeries; it has been used to provide intraoperative and postoperative analgesia.

The transversus abdominis plane is between the internal oblique muscle and the transversus abdominis muscle. In this plane, ilioinguinal and iliohypogastric nerves are located together. Ilioinguinal and iliohypogastric nerves originate from the ventral branches of L1 and in some variations, T12 may also contribute. The sensory innervation of the femoral region where endovascular cardiac interventions are performed is complex. It is thought that the ilioinguinal and iliohypogastric nerves contribute mostly. TAPB aims to provide analgesia by creating a block in these nerve branches that contribute to the sensory innervation of the intervention area.

ELIGIBILITY:
Inclusion Criteria:

* The patient is over 18 years of age
* Coronary angiography, cardiac catheterization and percutaneous coronary intervention will be applied to the patient,
* The above-mentioned procedures will be taken under elective conditions,
* Providing an optimal image when imaging the patient with ultrasound,
* INR< 1.5
* If the patient gives consent, S/he will be included in the study.

Exclusion Criteria:

* Patients under 18 years of age,
* Patients treated under emergency conditions,
* morbid obesity (BMI>35 kg/m2),
* pregnant women,
* New York Heart Association (NYHA) stage 4 patients with advanced decompensated heart failure,
* Patients with symptoms such as redness, temperature increase, infection, hematoma in the application area before the procedure,
* Patients with a history of allergy to local anesthetics,
* Patients who cannot be communicated,
* Those with severe psychosis or progressive neurological deficits and muscle disease,
* Patients who do not consent to the application will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
measuring the analgesic efficacy of TAPB | 4 months
  The pain will be assessed by the Numeric Rating Scale-11(NRS -11) to measure the analgesic efficacy of TAPB. Minimum pain score is point zero, maximum pain score is ten points.Minimum pain scores (NRS is less than 4 points) will have positive outcomes.
For patient and physician satisfaction;5-point Likert scale will be used. Minimum satisfaction score is one point, maksimum satisfaction score is five points.Higher scores have positive outcomes. | 4 months
  One point represents strongly unsatisfied and 5 points represent strongly satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Erkalp, Study Chair — Proffessor
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)